CLINICAL TRIAL: NCT06130059
Title: Pilot Study to Evaluate the Efficacy of Low Dose Colchicine (LoDoCo ®) to Improve Exercise Capacity Among Patients With Chronic Stable HFpEF and Systemic Inflammation
Brief Title: Efficacy of LoDoCo in Improving Exercise Capacity Among Patients With HFpEF and Inflammation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ambarish Pandey, Associate professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU-2023-0964
Record Dates: First submitted 2023-10-24; First posted 2023-11-13 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure; Inflammation
MeSH Terms: conditions — Heart Failure; Inflammation | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low dose colchicine (Experimental): Low dose colchicine 0.5 mg once a day orally for 3 months
  Interventions: Drug: Low Dose Colchicine
- Placebo (Placebo Comparator): Placebo once a day orally for 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low Dose Colchicine — Colchicine has been demonstrated to improve cardiovascular outcomes among patients with cardiovascular disease. In the COLCOT trial, the use of low-dose colchicine resulted in a reduction of major adverse cardiovascular events among participants with recent MI. The trial demonstrated the utility of anti-inflammatory therapies in improving cardiovascular outcomes. Colchicine has been widely used for decades and its safety profile is well established.
  Other Names: LoDoCo
  Arms: Low dose colchicine
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this research study is to determine the effectiveness of low dose colchicine (LoDoCo) on measures of exercise capacity, physical function, frailty, and quality of life, among patients with heart failure with chronic stable preserved ejection fraction (HFpEF) and systemic inflammation. The use of LoDoCo in this study is considered investigational as it has not been approved by the Food and Drug Administration (FDA) for the treatment of exercise capacity in patients with HFpEF.

Participants will undergo a 1-day screening that includes a blood draw and physical examination. If deemed eligible for the study, participants will undergo a baseline visit within 2 weeks of screening visit that includes physical examination, exercise testing, echocardiography and completion of quality-of-life surveys. Participants will also be randomized at this visit (randomly assigned to a group) to receive either LoDoCo or placebo (inactive substance) for 3 months. Participants will be called back at 3 months for repeat physical examination, blood draws, echocardiography, exercise testing and completion of quality-of-life surveys. Each visit will take about 3 hours. Total study duration is about 3 months.

DETAILED DESCRIPTION:
The investigators propose a single-center, double-blind placebo-controlled pilot study of LoDoCo vs. matching placebo among patients with chronic stable HFpEF and systemic inflammation. Patients that meet the eligibility criteria will be recruited prospectively from the UT Southwestern HFpEF program. Outcomes of interest will be assessed at baseline and 3 months. The primary outcome of the trial will be VO2peak indexed to body weight, and key secondary outcomes will include - 6MWD, KCCQ, change in structure and functional parameters of heart and hs-CRP levels.

Study Site:

UT Southwestern HFpEF program: The UT Southwestern HFpEF program, established in 2021 and is an integrated clinical and research enterprise that is responsible for the clinical care of patients with HFpEF and receives internal referrals from primary care, hospital medicine, geriatrics, and cardiology within the UT Southwestern health system and from clinics and hospitals in Texas and neighboring states. In the last year, the clinic has received over 300 referrals. The clinical program is integrated with an active research program that focuses on the phenotypic characterization of patients with HFpEF with an emphasis on exercise phenotyping. All patients with suspicion of HFpEF have a detailed laboratory, invasive hemodynamic, echocardiographic, and cardiopulmonary exercise testing. An active registry of patients is maintained which currently has ~150 participants with an established diagnosis of HFpEF and detailed phenotyping assessment.

The HFpEF clinic will serve as the clinical site of the study. Dr. Ambarish Pandey (PI) serves as the medical director of the HFpEF program.

Recruitment:

Detailed eligibility criteria are listed below. Participants will be drawn from the UT Southwestern HFpEF registry. The target enrollment for the study is 60 participants. Historical records and baseline evaluations will be used to determine eligibility for the study. After informed consent, participants will undergo study assessments as listed below followed by randomization.

Study Assessments (screening ):

Physical exam and vitals: Height, Weight and vitals - blood pressure, heart rate and SpO2 will be measured

Blood tests: Routine blood tests including creatinine, liver function tests, hemoglobin, hematocrit, serum chemistries, hs-CRP, and NT-proBNP. Blood assessments will be performed at the time of the baseline visit and 3-months post-treatment. (30 ml blood will be collected in the whole study)

Baseline and randomization (within 2 weeks of screening) Physical exam and vitals: Height, Weight and vitals - blood pressure, heart rate and SpO2 will be measured

Echocardiography: Echocardiography (ultrasound tests) of the heart before and after exercise and submaximal handgrip will be performed at baseline and follow-up. This is a non-invasive procedure in which the examination will be performed during supine rest to obtain standard two-dimensional images in the parasternal long and short axis and the apical two and four heart chamber views. To take pictures of patient's heart, a small non-invasive scanning probe with gel that will be applied to the participant's chest. Small adhesive pads will also be placed with wires to measure the participant's heart rate. It is anticipated that this procedure will not take more than 1 hour.

6-minute walking distance: The 6MWD assesses the distance a participant can walk in six minutes. It is a direct and timed measure of walking ability, which is technically simple, reproducible, and when administrators. are well trained, and readily standardized. The goal is for the subject to walk as far as possible in six minutes without running. The subject can self-pace and rest as needed as the subjects traverse back and forth along a marked walkway of 66 feet (20 m).

Kansas City Cardiomyopathy Questionnaire: (KCCQ): KCCQ measures Health-Related Quality of Life (HRQOL) and is a disease-specific health status instrument for HF. The approximate completion time is 4-6 minutes. Scores range from 0 to 100, with 0 as the lowest score and 100 as the highest score. Higher scores indicate better health status, fewer symptoms, and greater disease-specific health-related quality of life, respectively. The overall summary score and all domains have been independently demonstrated to be valid, reliable, and responsive to clinical change. The questionnaire consists of 23 items yielding:

7 domain scores (score range):

* Physical limitation (0-100)
* Symptom frequency (0-100)
* Symptom severity (0-100)
* Symptom stability (0-100)
* Self-efficacy and knowledge (0-100)
* Quality of life (0-100)
* Social limitation (0-100) 2 summary scores (score range):
* Total symptom score (0-100)
* Clinical summary score (CSS) (0-100) Overall summary score (score range: 0-100).

Cardiopulmonary Exercise testing: VO2peak, Participants will perform a maximal stress test on the upright cycle ergometer (Lode Corival CPET, Groningen, Netherlands). Participants will perform a continuous ramp protocol with a continuous increase in workload until maximal exhaustion. Respiratory gases including oxygen and carbon dioxide will be measured continuously using a metabolic cart (Ultima™ CardioO2 ® gas exchange analysis system; Saint Paul, Minnesota, USA) with measurements of expired oxygen and carbon dioxide and analyzed using Breeze Suit (Saint Paul, Minnesota, USA). The study team will determine maximal heart rate, peak oxygen uptake (VO2), carbon dioxide production (VCO2), pulmonary ventilation (VE), ventilatory equivalents for oxygen (VE/VO2), carbon dioxide (VE/CO2), respiratory exchange ratio (RER), end-tidal partial pressure of oxygen (PETO2), and carbon dioxide (PETCO2). Assessments will be performed at the time of the baseline visit, and 3 months post-treatment.

Randomization:

After review of baseline assessments. Qualifying Participants will be randomized to active study drug or matching placebo using a 1:1 block randomization scheme. The investigational drug service at UT Southwestern will store the study drug, perform randomization, and dispense the investigational product. Both participants and the study team will be blinded to treatment assignment.

3 months

Physical exam and vitals: Height, Weight and vitals - blood pressure, heart rate and SpO2 will be measured

Blood tests: Routine blood tests including creatinine, liver function tests, hemoglobin, hematocrit, serum chemistries, hs-CRP, and NT-proBNP. Blood assessments will be performed at the time of the baseline visit and 3-months post-treatment. (30 ml blood will be collected in the whole study)

Echocardiography: Echocardiography (ultrasound tests) of the heart before and after exercise and submaximal handgrip will be performed. This is a non-invasive procedure in which the examination will be performed during supine rest to obtain standard two-dimensional images in the parasternal long and short axis and the apical two and four heart chamber views. To take pictures of patient's heart, a small non-invasive scanning probe with gel that will be applied to the participant's chest. Small adhesive pads will also be placed with wires to measure the participant's heart rate. It is anticipated that this procedure will not take more than 1 hour.

6-minute walking distance: The 6MWD assesses the distance a participant can walk in six minutes. It is a direct and timed measure of walking ability, which is technically simple, reproducible, and when administrators. are well trained, and readily standardized. The goal is for the subject to walk as far as possible in six minutes without running. The subject can self-pace and rest as needed as the subjects traverse back and forth along a marked walkway of 66 feet (20 m).

Kansas City Cardiomyopathy Questionnaire: (KCCQ): KCCQ measures Health-Related Quality of Life (HRQOL) and is a disease-specific health status instrument for HF. The approximate completion time is 4-6 minutes. Scores range from 0 to 100, with 0 as the lowest score and 100 as the highest score. Higher scores indicate better health status, fewer symptoms, and greater disease-specific health-related quality of life, respectively. The overall summary score and all domains have been independently demonstrated to be valid, reliable, and responsive to clinical change. The questionnaire consists of 23 items yielding:

7 domain scores (score range):

* Physical limitation (0-100)
* Symptom frequency (0-100)
* Symptom severity (0-100)
* Symptom stability (0-100)
* Self-efficacy and knowledge (0-100)
* Quality of life (0-100)
* Social limitation (0-100) 2 summary scores (score range):
* Total symptom score (0-100)
* Clinical summary score (CSS) (0-100) Overall summary score (score range: 0-100).

Cardiopulmonary Exercise testing: VO2peak, Participants will perform a maximal stress test on the upright cycle ergometer (Lode Corival CPET, Groningen, Netherlands). Participants will perform a continuous ramp protocol with a continuous increase in workload until maximal exhaustion. Respiratory gases including oxygen and carbon dioxide will be measured continuously using a metabolic cart (Ultima™ CardioO2 ® gas exchange analysis system; Saint Paul, Minnesota, USA) with measurements of expired oxygen and carbon dioxide and analyzed using Breeze Suit (Saint Paul, Minnesota, USA). The study team will determine maximal heart rate, peak oxygen uptake (VO2), carbon dioxide production (VCO2), pulmonary ventilation (VE), ventilatory equivalents for oxygen (VE/VO2), carbon dioxide (VE/CO2), respiratory exchange ratio (RER), end-tidal partial pressure of oxygen (PETO2), and carbon dioxide (PETCO2). Assessments will be performed at the time of the baseline visit, and 3 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Informed consent was obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.

  2. Age 50 years or above at the time of signing the informed consent. 3. Serum hs-CRP 2 mg/L at the time of baseline testing. 4. Diagnosis of chronic HFpEF within 6 months of enrolment must have one of the following:

  a. Structural Heart Disease with one of the following on echocardiography within 12 months of enrolment.

  i. LA volume index > 34 ml/m2. ii. LA diameter ≥ 3.8 cm. iii. LA length ≥ 5.0 cm. iv. LA area ≥ 20 cm2. v. LA volume ≥ 55 mL. vi. Intraventricular septal thickness ≥1.1 cm. vii. Posterior wall thickness ≥1.1 cm. viii. LV mass index ≥115 g∕m2 in men or ≥ 95 g∕m2 in women. ix. E/e' (mean septal and lateral) ≥ 10. x. e' (mean septal and lateral) < 9 cm/s b. Pulmonary capillary wedge pressure (PCWP) at rest³15 mmHg or Left ventricular end-diastolic pressure (LVEDP) ³18 mmHg, (PCWP) with exercise ³25 mmHg or (³ 2 mmHg/L/min) c. HF hospitalization or urgent/unplanned visit with a primary diagnosis of decompensated heart failure which required intravenous loop diuretic treatment, within the last 9 months prior to enrolment in combination with NT-proBNP ≥ 125 pg/mL within 1 month of enrolment for patients without ongoing atrial fibrillation/flutter. If ongoing atrial fibrillation/flutter at screening NT-proBNP must be ≥ 300 pg/mL 5. Ambulatory participants who can perform cardiopulmonary exercise testing. 6. Stable doses of HF-specific medications within the last 1 month. 7. Stable level of physical activity 8. Stable dose of any weight loss medications.

Exclusion Criteria:

* 1. Do not otherwise meet the inclusion criteria. 2. Women who are pregnant, breastfeeding, or may be considering pregnancy during the study period.

  3. Renal impairment: eGFR <30mL/min 4. Severe valvular heart disease is considered likely to require intervention. 5. Life expectancy <1 year. 6. Unable to perform cardiopulmonary exercise testing. 7. ALT or AST >2.5 ULN at time of screening

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Peak VO2 indexed to body weight | Over 3 months
  The primary outcome of the trial will be VO2peak indexed to body weight. (mL/kg/min). The data will be analyzed on an intention-to-treat basis comparing the outcomes across treatment arms (LoDoCo vs. placebo) using analysis of variance for repeated measures (ANOVA). Randomization of 60 participants (30 in LoDoCo vs. placebo) will provide >80% power at a two-sided level of significance of 0.05 to detect a >15% difference in VO2peak at the end of the study period. This estimate assumes a target population mean VO2peak of 10.5 ml/kg/min (SD 2.9) based on data from our local registry. Assuming a dropout rate of ~20%, we will plan to enroll 72 participants. We will also evaluate the association between changes in hs-CRP with changes in VO2peak across the entire cohort of participants using adjusted linear and logistic regression models

SECONDARY OUTCOMES:
Difference in 6 minute walk distance | 3 months
  It will be assessed using analysis of covariance (ANCOVA). The randomized arm will be the between-subject grouping variable; covariates will be baseline value, baseline age, sex, and hs-CRP. The least-square means will be used to estimate intervention effects. Tests will be conducted at the 5% two-sided level of significance. The appropriate transformation will be used for biomarkers with skewed distributions to stabilize variance and achieve better approximation to normality.
Difference in Kansas City Cardiomyopathy Questionnaire - Clinical Summary Score (KCCQ) Score | 3 months
  It will be assessed using analysis of covariance (ANCOVA). The randomized arm will be the between-subject grouping variable; covariates will be baseline value, baseline age, sex, and hs-CRP. The least-square means will be used to estimate intervention effects. Tests will be conducted at the 5% two-sided level of significance. The appropriate transformation will be used for biomarkers with skewed distributions to stabilize variance and achieve better approximation to normality. Scores range from 0 to 100, with 0 as the lowest score and 100 as the highest score. Higher scores indicate better health status, fewer symptoms, and greater disease-specific health-related quality of life, respectively.
Percent change cardiac structure and function | Baseline and 3 months
  Echocardiography at baseline and follow-up will be used to determine changes in cardiac structure and function. Left atrial, and ventricular sizes will be measured at end-diastole and end-systole. Cardiac systolic function will be measured using left ventricular ejection fraction. Diastolic function will be measured as tissue Doppler velocities - E/e', and e' velocities. Absolute, and percent changes in these parameters between baseline and follow-up will be measured as an exploratory outcome. Analysis of covariance (ANCOVA) will be used for the analysis of the effect of the intervention. The randomized arm will be the between-subject grouping variable; covariates will be baseline value, baseline age, sex The least-square means will be used to estimate intervention effects.
Difference in hs-CRP levels | 3 months
  It will be assessed using analysis of covariance (ANCOVA). The randomized arm will be the between-subject grouping variable; covariates will be baseline value, baseline age, sex, and hs-CRP. The least-square means will be used to estimate intervention effects. Tests will be conducted at the 5% two-sided level of significance. The appropriate transformation will be used for biomarkers with skewed distributions to stabilize variance and achieve better approximation to normality.

CONTACTS AND LOCATIONS:
Overall Officials: Ambarish Pandey, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW; ACC/AHA Joint Committee Members. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2022 May 3;145(18):e895-e1032. doi: 10.1161/CIR.0000000000001063. Epub 2022 Apr 1. PMID 35363499
- [Background] Nayor M, Houstis NE, Namasivayam M, Rouvina J, Hardin C, Shah RV, Ho JE, Malhotra R, Lewis GD. Impaired Exercise Tolerance in Heart Failure With Preserved Ejection Fraction: Quantification of Multiorgan System Reserve Capacity. JACC Heart Fail. 2020 Aug;8(8):605-617. doi: 10.1016/j.jchf.2020.03.008. Epub 2020 Jun 10. PMID 32535122
- [Background] Pandey A, Shah SJ, Butler J, Kellogg DL Jr, Lewis GD, Forman DE, Mentz RJ, Borlaug BA, Simon MA, Chirinos JA, Fielding RA, Volpi E, Molina AJA, Haykowsky MJ, Sam F, Goodpaster BH, Bertoni AG, Justice JN, White JP, Ding J, Hummel SL, LeBrasseur NK, Taffet GE, Pipinos II, Kitzman D. Exercise Intolerance in Older Adults With Heart Failure With Preserved Ejection Fraction: JACC State-of-the-Art Review. J Am Coll Cardiol. 2021 Sep 14;78(11):1166-1187. doi: 10.1016/j.jacc.2021.07.014. PMID 34503685
- [Background] Kalogeropoulos A, Georgiopoulou V, Psaty BM, Rodondi N, Smith AL, Harrison DG, Liu Y, Hoffmann U, Bauer DC, Newman AB, Kritchevsky SB, Harris TB, Butler J; Health ABC Study Investigators. Inflammatory markers and incident heart failure risk in older adults: the Health ABC (Health, Aging, and Body Composition) study. J Am Coll Cardiol. 2010 May 11;55(19):2129-37. doi: 10.1016/j.jacc.2009.12.045. PMID 20447537
- [Background] Schiattarella GG, Altamirano F, Tong D, French KM, Villalobos E, Kim SY, Luo X, Jiang N, May HI, Wang ZV, Hill TM, Mammen PPA, Huang J, Lee DI, Hahn VS, Sharma K, Kass DA, Lavandero S, Gillette TG, Hill JA. Nitrosative stress drives heart failure with preserved ejection fraction. Nature. 2019 Apr;568(7752):351-356. doi: 10.1038/s41586-019-1100-z. Epub 2019 Apr 10. PMID 30971818
- [Background] Franssen C, Chen S, Unger A, Korkmaz HI, De Keulenaer GW, Tschope C, Leite-Moreira AF, Musters R, Niessen HW, Linke WA, Paulus WJ, Hamdani N. Myocardial Microvascular Inflammatory Endothelial Activation in Heart Failure With Preserved Ejection Fraction. JACC Heart Fail. 2016 Apr;4(4):312-24. doi: 10.1016/j.jchf.2015.10.007. Epub 2015 Dec 9. PMID 26682792
- [Background] Westermann D, Lindner D, Kasner M, Zietsch C, Savvatis K, Escher F, von Schlippenbach J, Skurk C, Steendijk P, Riad A, Poller W, Schultheiss HP, Tschope C. Cardiac inflammation contributes to changes in the extracellular matrix in patients with heart failure and normal ejection fraction. Circ Heart Fail. 2011 Jan;4(1):44-52. doi: 10.1161/CIRCHEARTFAILURE.109.931451. Epub 2010 Nov 12. PMID 21075869
- [Background] DuBrock HM, AbouEzzeddine OF, Redfield MM. High-sensitivity C-reactive protein in heart failure with preserved ejection fraction. PLoS One. 2018 Aug 16;13(8):e0201836. doi: 10.1371/journal.pone.0201836. eCollection 2018. PMID 30114262
- [Background] Tromp J, Khan MA, Klip IT, Meyer S, de Boer RA, Jaarsma T, Hillege H, van Veldhuisen DJ, van der Meer P, Voors AA. Biomarker Profiles in Heart Failure Patients With Preserved and Reduced Ejection Fraction. J Am Heart Assoc. 2017 Mar 30;6(4):e003989. doi: 10.1161/JAHA.116.003989. PMID 28360225
- [Background] Hage C, Michaelsson E, Linde C, Donal E, Daubert JC, Gan LM, Lund LH. Inflammatory Biomarkers Predict Heart Failure Severity and Prognosis in Patients With Heart Failure With Preserved Ejection Fraction: A Holistic Proteomic Approach. Circ Cardiovasc Genet. 2017 Feb;10(1):e001633. doi: 10.1161/CIRCGENETICS.116.001633. PMID 28100627
- [Background] Kitzman DW, Haykowsky MJ, Tomczak CR. Making the Case for Skeletal Muscle Myopathy and Its Contribution to Exercise Intolerance in Heart Failure With Preserved Ejection Fraction. Circ Heart Fail. 2017 Jul;10(7):e004281. doi: 10.1161/CIRCHEARTFAILURE.117.004281. No abstract available. PMID 28705911
- [Background] Fleg JL, Cooper LS, Borlaug BA, Haykowsky MJ, Kraus WE, Levine BD, Pfeffer MA, Pina IL, Poole DC, Reeves GR, Whellan DJ, Kitzman DW; National Heart, Lung, and Blood Institute Working Group. Exercise training as therapy for heart failure: current status and future directions. Circ Heart Fail. 2015 Jan;8(1):209-20. doi: 10.1161/CIRCHEARTFAILURE.113.001420. No abstract available. PMID 25605639
- [Background] Warraich HJ, Kitzman DW, Whellan DJ, Duncan PW, Mentz RJ, Pastva AM, Nelson MB, Upadhya B, Reeves GR. Physical Function, Frailty, Cognition, Depression, and Quality of Life in Hospitalized Adults >/=60 Years With Acute Decompensated Heart Failure With Preserved Versus Reduced Ejection Fraction. Circ Heart Fail. 2018 Nov;11(11):e005254. doi: 10.1161/CIRCHEARTFAILURE.118.005254. PMID 30571197
- [Background] Chiarantini D, Volpato S, Sioulis F, Bartalucci F, Del Bianco L, Mangani I, Pepe G, Tarantini F, Berni A, Marchionni N, Di Bari M. Lower extremity performance measures predict long-term prognosis in older patients hospitalized for heart failure. J Card Fail. 2010 May;16(5):390-5. doi: 10.1016/j.cardfail.2010.01.004. Epub 2010 Mar 3. PMID 20447574
- [Background] Pandey A, Kitzman D, Whellan DJ, Duncan PW, Mentz RJ, Pastva AM, Nelson MB, Upadhya B, Chen H, Reeves GR. Frailty Among Older Decompensated Heart Failure Patients: Prevalence, Association With Patient-Centered Outcomes, and Efficient Detection Methods. JACC Heart Fail. 2019 Dec;7(12):1079-1088. doi: 10.1016/j.jchf.2019.10.003. PMID 31779931
- [Background] Murad K, Goff DC Jr, Morgan TM, Burke GL, Bartz TM, Kizer JR, Chaudhry SI, Gottdiener JS, Kitzman DW. Burden of Comorbidities and Functional and Cognitive Impairments in Elderly Patients at the Initial Diagnosis of Heart Failure and Their Impact on Total Mortality: The Cardiovascular Health Study. JACC Heart Fail. 2015 Jul;3(7):542-550. doi: 10.1016/j.jchf.2015.03.004. PMID 26160370
- [Background] Ather S, Chan W, Bozkurt B, Aguilar D, Ramasubbu K, Zachariah AA, Wehrens XH, Deswal A. Impact of noncardiac comorbidities on morbidity and mortality in a predominantly male population with heart failure and preserved versus reduced ejection fraction. J Am Coll Cardiol. 2012 Mar 13;59(11):998-1005. doi: 10.1016/j.jacc.2011.11.040. PMID 22402071
- [Background] Kitzman DW, Brubaker P, Morgan T, Haykowsky M, Hundley G, Kraus WE, Eggebeen J, Nicklas BJ. Effect of Caloric Restriction or Aerobic Exercise Training on Peak Oxygen Consumption and Quality of Life in Obese Older Patients With Heart Failure With Preserved Ejection Fraction: A Randomized Clinical Trial. JAMA. 2016 Jan 5;315(1):36-46. doi: 10.1001/jama.2015.17346. PMID 26746456
- [Background] Van Tassell BW, Buckley LF, Carbone S, Trankle CR, Canada JM, Dixon DL, Abouzaki N, Oddi-Erdle C, Biondi-Zoccai G, Arena R, Abbate A. Interleukin-1 blockade in heart failure with preserved ejection fraction: rationale and design of the Diastolic Heart Failure Anakinra Response Trial 2 (D-HART2). Clin Cardiol. 2017 Sep;40(9):626-632. doi: 10.1002/clc.22719. Epub 2017 May 5. PMID 28475816
- [Background] Tardif JC, Kouz S, Waters DD, Bertrand OF, Diaz R, Maggioni AP, Pinto FJ, Ibrahim R, Gamra H, Kiwan GS, Berry C, Lopez-Sendon J, Ostadal P, Koenig W, Angoulvant D, Gregoire JC, Lavoie MA, Dube MP, Rhainds D, Provencher M, Blondeau L, Orfanos A, L'Allier PL, Guertin MC, Roubille F. Efficacy and Safety of Low-Dose Colchicine after Myocardial Infarction. N Engl J Med. 2019 Dec 26;381(26):2497-2505. doi: 10.1056/NEJMoa1912388. Epub 2019 Nov 16. PMID 31733140